CLINICAL TRIAL: NCT03040063
Title: Complex Endovascular Approach to Treatment of Patients With Aneurysm of Popliteal Artery and Acute Limb Ischemia
Brief Title: Complex Endovascular Approach to Treatment of Patients With Aneurysm of Popliteal Artery
Acronym: EVAR-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Petr Varejka (Unknown)
Responsible Party: Principal Investigator, Ass. prof. Jean-Claude M. Lubanda, MD, Ph.D, Ass.prof. MD, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVAR-P
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Aneurysm; Popliteal Artery; Limb Ischemia
Keywords: aneurysm, poplietl artery, acute limb ischemia
MeSH Terms: conditions — Popliteal Artery Aneurysm; Aneurysm

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined endovascular approach (Experimental): Combined endovascular approach using covered stent and flexible stent in the popliteal artery
  Interventions: Procedure: Combined endovascular approach (EVAR)
- Standard optimal therapy (OPT) (Experimental): standard therapy of popliteal artery aneurysm using thrombolysis and surgery
  Interventions: Procedure: Standard optimal therapy (OPT)

INTERVENTIONS:
Procedure: Combined endovascular approach (EVAR) — 1. puncture of SFA in orthograde position if possible
  2. DSA through 4F dilator, proof of occlusion
  3. wire test
  4. Heparin 70-80 IU/kg i.a.
  5. implantation of peripheral stent graft VIABAHN
  6. implantation of peripheral stent SUPERA into stent graft
  7. insertion of strait flush catheter for local thrombolysis
  8. administration of continuous local thrombolysis in the dose of 1 mg/hr., unfractionated heparin continuously (APTT 1,5-2x) according to the department standards
  9. control angiography in 12 hrs or earlier according to clinical status and symptoms
  10. repeated angiography in 24 hrs
  Arms: Combined endovascular approach
Procedure: Standard optimal therapy (OPT) — 1. puncture of SFA in orthograde position if possible
  2. DSA through 4F dilator, proof of occlusion
  3. wire test
  4. Unfractionated heparin 70-80 IU/kg i.a.
  5. insertion of strait flush catheter for local thrombolysis
  6. administration of continuous local thrombolysis in the dose of 1 mg/hr., unfractionated heparin continuously (APTTT 1,5-2x)
  7. control angiography in 12 hrs or according to clinical status and symptoms
  8. repeated angiography in24 hrs
  9. Final result review, vascular team consultation and indication for surgical or conservative management of popliteal artery aneurysm.
  Arms: Standard optimal therapy (OPT)

SUMMARY:
Use of endovascular techniques - implantation of a peripheral stent graft and a peripheral flexible stent to isolate the sac of the popliteal artery aneurysm from the circulation and subsequent topical application of a thrombolytic (rtPA) to restore patency of the lower leg blood stream - will lead to a comparable or better outcome in treatment of patients with the popliteal artery aneurysm and acute critical limb ischaemia, compared to currently prevailing use of surgical treatment.

DETAILED DESCRIPTION:
The 2nd Medical Department admits patients with acute arterial occlusion at the stage of critical limb ischaemia. The poorest prognosis considering preservation of the limb is shown by the patients who exhibit symptoms of ischaemia due to affected popliteal artery and arteries of the shank in the the popliteal artery aneurysm. On the other hand, diagnosis of this condition is prompt and easy (general ultrasound scan below the knee). Patients with the popliteal artery aneurysm, confirmed by ultrasound investigation, and concurrent signs and symptoms of acute critical ischaemia will be indicated for catheterization intervention at our unit, which will confirm morphological compatibility with endovascular occlusion of the aneurysm sac through implantation of a peripheral stent graft, supported by implantation of a peripheral flexible stent, and at the same time insertion of a thrombolytic catheter into the implanted stent graft for local thrombolysis of tibial arteries if required by the current situation. The patient will be hospitalized at the angiology intensive care unit of the 2nd Medical Department, where local intra-arterial thrombolytic therapy will be performed according to the standard protocol. After completion of the proper endovascular treatment, the patients will be transferred to combined peroral anticoagulation and antiaggregation treatment, and all of them will have an ultrasound scan below the knee, with the readings archived for the purpose of further comparison and monitoring. Subsequently, the patients will be monitored in the outpatient regime after 6 weeks, 3, 6 and 12 months. At each visit, clinical examination will be done including establishment of ABI/TBI values and ultrasound investigation of the region below the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form for the patient's participation in the study.
2. Acute critical limb ischaemia with impairment of the extremity at stage I, IIa, IIb according to SVS classification.
3. A popliteal artery aneurysm, confirmed by ultrasound scanning, which on catheterization examination meets the criteria for isolation of the aneurysm sac by implantation of a peripheral stent graft, supported by insertion of a peripheral flexible stent.
4. Absence of any contraindication for local thrombolytic therapy.
5. An anatomic finding through angiographic investigation that is suitable for endovascular therapy.

Exclusion Criteria:

1. Active bleeding or contraindication for local thrombolysis.
2. Life expectance < 1 yr
3. Relevant stenotic defects of valves.
4. Myocardial infarction or unstable angina pectoris in past 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Limb salvage in 12 months | 12 Months
  Limba salvage in 12 months
Patency of the popliteal artery in 12 months | 12 Months
  Patency of the popliteal artery in 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charles University in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No